CLINICAL TRIAL: NCT07196020
Title: Prediction and Prevention of Venous Thrombo-embolism(VTE) During Chemotherapy Using Serial Determination of Haemostasis Biomarkers.
Brief Title: Prediction of Venous Thrombosis During chemotherapy-the PINPOINT Study
Acronym: PINPOINT
Status: Not yet recruiting | Type: Observational
Sponsor: University of Dublin, Trinity College (Other)
Collaborators: Cork University Hospital (Other); Mater Misericordiae University Hospital (Other)
Responsible Party: Principal Investigator, Lucy Norris, Principal Investigator/Research Fellow, University of Dublin, Trinity College
Other Study IDs: ILP-POR-2024-029
Record Dates: First submitted 2025-09-18; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Venous Thromboembolism; Cancer
Keywords: Chemotherapy; Cancer; Thrombin; Venous thromboembolism; Neoplasms
MeSH Terms: conditions — Venous Thromboembolism; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma samples (citrated plasma)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cancer patients undergoing chemotherapy: Lung, ovarian and pancreatic cancer patients undergoing chemotherapy.

SUMMARY:
Cancer patients are at higher risk of getting a blood clot (known as venous thromboembolism (VTE)) especially during chemotherapy and some patients are more at risk than others. These clots can be prevented by using blood thinners (known as anticoagulants) but these are not suitable for everyone as they also carry a risk of bleeding. This study aims to identify which chemotherapy patients are most at risk of a blood clot and at what point in their treatment this is likely to happen. In this project biomarkers in the blood that are involved in blood clotting will be measured in cancer patients at four stages during chemotherapy to see how the biomarkers change during treatment. The blood samples for these tests are taken at the same time as the normal routine blood tests done before a chemotherapy cycle. Biomarker levels will be compared between those patients who subsequently get a VTE and those who do not get a VTE. This will help develop a biomarker based blood test to predict clots during chemotherapy. The biomarker based test will also be compared with other methods of predicting VTE in cancer patients which are currently in use. In the future, this blood test might be used to see if patients are at high risk of a clot during chemotherapy and provide a method to optimise the use of preventative anticoagulants in cancer patients during chemotherapy.

DETAILED DESCRIPTION:
Background:

VTE is the leading cause of death in cancer patients after the cancer itself. Amongst solid tumours, pancreatic, lung, brain, stomach, and ovarian cancer are the most prothrombotic and are associated with high rates of VTE depending on tumour histology and treatment. The recommended tool for VTE risk assessment during chemotherapy is the Khorana risk score, which was designed to identify ambulatory cancer patients at increased risk of VTE during chemotherapy. This tool has been recommended for use in guiding thromboprophylaxis in cancer patients undergoing chemotherapy. However, the Khorana score performs poorly in cancers of a single type, especially cancers at high risk of VTE. Previous studies have used a variety of biomarkers to predict VTE in cancer patients, however prediction was based on one sample and does not account for the dynamic nature of thrombogenesis particularly during chemotherapy. Dynamic risk assessment using serial measurement of biomarkers during therapy has been recommended as a more effective approach to risk assessment. Guidelines have suggested repeated risk assessment using the new Vienna CAT score (a nomogram based on D-dimer levels and tumour site) may improve risk prediction. Preliminary data has shown suggests that three novel biomarkers may be (soluble Thrombomodulin(TM), Thrombin generation assay[TGA] and Factor VIIIc (FVIIIc) levels) measured serially may be effective alone or in combination as dynamic predictive biomarkers for VTE during chemotherapy.

Study objective:

The aim of the study is to measure these three biomarkers (TGA, TM and FVIIIc) serially in lung, ovarian, pancreatic and gastric cancer patients undergoing chemotherapy to dynamically assess the ability of these biomarkers to predict VTE.

Study Design:

The study will recruit 380 patients across three centres in Ireland. Blood samples will be taken from each patient at the following stages during chemotherapy treatment.

1. Before chemotherapy treatment
2. after 4 weeks treatment
3. after 3 months treatment
4. at the end of the current cycle of treatment.

Based on clinical data available, the Khorana Risk Score(KRS) calculated at the start of therapy. The Vienna CAT nomogram will be calculated at each sampling point in the study.

Laboratory Biomarker analysis:

All biomarker analysis will take place at the Coagulation Research Laboratory, Dept of Obstetrics and Gynaecology, Trinity St. James Cancer Institute, St. James's Hospital. Dublin IRELAND sTM will be measured using Enzyme Linked Immunosorbent Assay (ELISA) and FVIIIc will be measured using chromogenic substrate assay . TGA will be measured using fluorimetric assay. D-dimer (for calculation of the Vienna CAT score) will be measured using a 2-step procedure.

All VTE events which occur from baseline to within 3 months of the final sample will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of ovarian, lung, gastric or pancreatic cancer scheduled to undergo a course of chemotherapy who are undergoing adjuvant or neoadjuvant chemotherapy, or who are undergoing chemotherapy for relapsed disease or patients receiving targeted therapy in combination with chemotherapy
* Patients who are over 18 years of age
* Patients who are able to give full and informed written consent

Exclusion Criteria:

* Prior history of a documented VTE event within the last 5 years (excluding central line associated events whereby patients completed anticoagulation > 3 months previously)
* Any history of significant haemorrhage (requiring hospitalization or transfusion) outside of a surgical setting within the last 5 years
* Familial bleeding diathesis
* Known diagnosis of disseminated intravascular coagulation.
* Surgery within 2 weeks of first baseline sample (with the exception of porth-a-cath implantation or biopsy)
* Chemotherapy or immunotherapy 4 weeks before first baseline sample
* Currently receiving long term anticoagulant therapy (Low Molecular Weight Heparin(LMWH), Direct Oral Anticoagulants(DOACs), Warfarin). Patients receiving aspirin, ticlopidine, clopidogrel or LMWH at a prophylactic dosage for a short period (ie post cancer surgery or during short hospital stay) will be included provided they have completed thromboprophylaxis therapy at the first blood sampling time point.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of ovarian, lung, gastric or pancreatic cancer who are scheduled to undergo a course of chemotherapy in the three study centres in Ireland.
Sampling Method: Non-Probability Sample
Enrollment: 380 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2029-03-01 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
Venous thromboembolism | From initiation of treatment to 12 weeks from last sample time point
  Venous thromboembolism during the chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Lucy A Norris, PhD, Principal Investigator — Trinity College Dublin (The University of Dublin, Ireland)
Locations (3):
- Ireland (3):
  - Cork University Hospital, Cork
  - Mater Misericordiae University Hospital, Dublin
  - Trinity Cancer St. James Cancer Institute, Dublin

IPD SHARING:
Plan to Share IPD: Undecided
Limitations according to GDPR regulations in Ireland on what can or cannot be shared

REFERENCES:
- [Background] Ward MP, Ibrahim EM, O'Toole SA, Marchocki Z, O'Leary JJ, Saadeh FA, Norris LA. Chemotherapy alters thrombomodulin and factor VIIIc expression resulting in acquired activated protein C resistance and enhanced thrombin generation in cancer associated thrombosis. Thromb Res. 2025 Feb;246:109251. doi: 10.1016/j.thromres.2024.109251. Epub 2024 Dec 30. PMID 39793535
- [Background] Pabinger I, van Es N, Heinze G, Posch F, Riedl J, Reitter EM, Di Nisio M, Cesarman-Maus G, Kraaijpoel N, Zielinski CC, Buller HR, Ay C. A clinical prediction model for cancer-associated venous thromboembolism: a development and validation study in two independent prospective cohorts. Lancet Haematol. 2018 Jul;5(7):e289-e298. doi: 10.1016/S2352-3026(18)30063-2. Epub 2018 Jun 7. PMID 29885940
- [Background] Khorana AA, Kuderer NM, Culakova E, Lyman GH, Francis CW. Development and validation of a predictive model for chemotherapy-associated thrombosis. Blood. 2008 May 15;111(10):4902-7. doi: 10.1182/blood-2007-10-116327. Epub 2008 Jan 23. PMID 18216292

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-03-15): https://cdn.clinicaltrials.gov/large-docs/20/NCT07196020/Prot_SAP_000.pdf
  • Informed Consent Form (2025-05-01): https://cdn.clinicaltrials.gov/large-docs/20/NCT07196020/ICF_001.pdf